CLINICAL TRIAL: NCT04048499
Title: Prevalence and Severity of Colour Vision Deficiency Among Turkish Children
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Funda Dikkaya, asist proffesor, Medipol University
Other Study IDs: 425
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: CAD Test; Children's Vision; Colour Assessment; Colour Vision; Turkey
MeSH Terms: interventions — Diagnosis; Diagnosis, Computer-Assisted

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: the Colour Assessment and Diagnosis (CAD) test — The CAD test (City Occupational Ltd, London, UK) measures the severity of red-green and yellow-blue colour vision loss according to red-green and yellow-blue thresholds which are expressed in CAD units and diagnoses accurately the subject's class of colour vision

SUMMARY:
To evaluate the usability of the Colour Assessment and Diagnosis (CAD) test in children. To determine the prevalence of colour vision deficiency (CVD) among Turkish children, to identify the class of deficiency and to quanify severity of loss.

ELIGIBILITY:
Inclusion Criteria: children with aged 6-16 years, who attended the ophthalmology department at the Istanbul Medipol University -

Exclusion Criteria:Children with known or current evidence of ocular pathology (other than refractive errors), with history of long term use of medication, previous ocular surgery and those with chronic systemic diseases were excluded from the study

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A total of 1374 children, aged 6-16 years, who attended the ophthalmology department at the Istanbul Medipol University were included in the study.
Sampling Method: Probability Sample
Enrollment: 1374 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Prevalence and Severity of Colour Vision Deficiency among Turkish Children | january 2018-march 2019
  number of children with colour vision deficiency (CVD) among Turkish children who attend to the clinic in a period o time, number of children in each class of deficiency (protan, deutan) and number of children in each category according to severity.
the usability of the Colour Assessment and Diagnosis (CAD) test in children | january 2018-march 2019
  number of children who were cooperative and carried out the full CAD test

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No